CLINICAL TRIAL: NCT01562145
Title: Elevated Plasma Levels of TIMP-1 in Patients With Rotator Cuff Tear
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Hanna Bjornsson, MD, Shoulder surgeon and head of shoulder research team, University Hospital, Linkoeping
Other Study IDs: HannaBjornssonstud3
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff tear, matrix metalloproteinase, tissue inhibitor of matrix metalloproteinase, partial-thickness tear, full-thickness tear, plasma.
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with rotator cuff tears: Patients with ultrasound verified rotator cuff tears
  Interventions: Procedure: Blood sampling
- Healthy controls: Age and gender matched controls with ultrasound verified intact rotator cuff
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Four mL venous blood samples were collected from all study participants after inclusion

SUMMARY:
The aim of the study was to investigate the levels of matrixmetalloproteinases and their inhibitors in blood samples from patients with rotator cuff tears and compare with blood samples from healthy matched controls.

DETAILED DESCRIPTION:
Background: Extracellular matrix remodeling is altered in rotator cuff tears, partly due to altered expression of matrix metalloproteinases (MMPs) and their inhibitors. It is unclear if this altered expression can be traced as changes in plasma protein levels. We measured the plasma level of MMPs and their tissue inhibitors (TIMPs) in patients with rotator cuff tears.

Material and methods: Blood samples were collected from 17 patients, median 61 (range 39-77) years, with sonographically verified rotator cuff tears (partial- or full-thickness). These were compared with 16 gender and age matched control persons with sonographically intact rotator cuffs. Plasma levels of MMPs and TIMPs were measured simultaneously using Luminex technology.

ELIGIBILITY:
Inclusion Criteria:

- degenerative rotator cuff tear verified by ultrasound

Exclusion Criteria:

* systemic joint disease such as rheumatoid arthritis
* a fracture non-union
* dupuytrens disease
* frozen shoulder
* tendinosis or rupture of any other tendons than in the rotator cuff
* disorders of the spine such as disc disease,idiopathic scoliosis, spondylitis
* cerebral or cardiovascular disease during the past year
* abdominal or bowel disease
* surgery or trauma during the past year
* any infection during the last month
* malignancy
* treatment for the last month with medications that may affect MMPs or TIMPs (tetracycline, bisphosphonates, anti-inflammatory drugs, statins)
* vigorous physical activity during the last 24 hours
* inability to understand written and spoken Swedish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ultrasound verified rotator cuff tears and healthy age and gender matched controls
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Level of MMP and TIMP in plasma | Measaured at one time point
  Four mL venous blood samples were collected from all study participants after inclusion, and centrifuged to plasma that was stored at -70 degrees until the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Björnsson Hallgren, MD, Principal Investigator — University clinic of orthopeadics Linkoeping
Locations (1):
- University clinic of orthopeadics Linkoeping, Linköping, Östergötland County, Sweden

REFERENCES:
- [Result] Pasternak B, Aspenberg P. Metalloproteinases and their inhibitors-diagnostic and therapeutic opportunities in orthopedics. Acta Orthop. 2009 Dec;80(6):693-703. doi: 10.3109/17453670903448257. PMID 19968600
- [Result] Lo IK, Marchuk LL, Hollinshead R, Hart DA, Frank CB. Matrix metalloproteinase and tissue inhibitor of matrix metalloproteinase mRNA levels are specifically altered in torn rotator cuff tendons. Am J Sports Med. 2004 Jul-Aug;32(5):1223-9. doi: 10.1177/0363546503262200. Epub 2004 May 18. PMID 15262646